CLINICAL TRIAL: NCT01153386
Title: An Evaluation of the Pharmacokinetic Linearity and Comparative Bioavailability of a Single Oral Dose of 0.5 mg, 1 mg and 2.5 mg UT-15C (Treprostinil Diethanolamine) SR Tablets in Healthy Volunteers in the Fed State
Brief Title: Pharmacokinetic Linearity and Comparative Bioavailability of Treprostinil Diethanolamine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Allison Lim, United Therapeutics
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TDE-PH-122
Record Dates: First submitted 2010-06-28; First posted 2010-06-30 (Estimated); Last update posted 2010-08-23 (Estimated); Status verified 2010-08

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary arterial hypertension; Treprostinil; Pharmacokinetics
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.5 mg treprostinil diethanolamine (Experimental): 0.5 mg treprostinil diethanolamine
  Interventions: Drug: Treprostinil diethanolamine
- 2.5 mg treprostinil diethanolamine (Experimental): 2.5 mg treprostinil diethanolamine
  Interventions: Drug: Treprostinil diethanolamine
- 1 mg treprostinil diethanolamine (Experimental): 1 mg treprostinil diethanolamine
  Interventions: Drug: Treprostinil diethanolamine

INTERVENTIONS:
Drug: Treprostinil diethanolamine — Treprostinil diethanolamine sustained release oral tablets.
  Other Names: UT-15C

SUMMARY:
This study will compare the bioavailability and pharmacokinetics of the 0.5 mg, 1 mg and 2.5 mg treprostinil diethanolamine tablet strengths in healthy volunteers.

DETAILED DESCRIPTION:
This study was designed to assess the pharmacokinetic linearity and comparative bioavailability of UT-15C SR (treprostinil diethanolamine) following the administration of a single tablet containing 0.5 mg, 1 mg and 2.5 mg UT-15C in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subject is healthy and between the ages of 18 and 55 years
* Female subjects must weigh between 55 and 100 kg, inclusive, with a BMI between 19.0-29.9 kg/m2, inclusive at Screening. Male subjects must weigh between 55 and 120 kg, inclusive, with a BMI between 19.0-32.0 kg/m2, inclusive at Screening.
* Subject has a medical history, physical examination, vital signs, ECG and clinical laboratory results within normal limits or considered not clinically significant by the Investigator at Screening.

Exclusion Criteria:

* Subject has any clinically relevant abnormality identified during the screening physical examination, 12-lead ECG, or laboratory examinations.
* Subject has a history of anaphylaxis, a documented hypersensitivity reaction, or a clinically significant idiosyncratic reaction to any drug.
* Subject has a clinically significant history of neurological, cardiovascular, respiratory, endocrine, hematological, hepatic, renal, gastrointestinal, genitourinary, pulmonary and/or musculoskeletal disease; glaucoma; a psychiatric disorder or any other chronic disease, whether controlled by medication or not.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Treprostinil pharmacokinetics | 36 hours
  Treprostinil pharmacokinetics in healthy volunteers following a single oral dose of 0.5 mg, 1 mg and 2.5 mg treprostinil diethanolamine sustained release tablets immediately prior to through 36 hours post treprostinil diethanolamine dosing.

SECONDARY OUTCOMES:
Clinical laboratories | Study Days 0, 7, 14 and 16.
Adverse event monitoring | From the first dose of treprostinil diethanolamine through the end of the study (Study Day 16)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Hunt, MD, PhD, Principal Investigator — PPD Development, LP
Locations (1):
- PPD Development, Austin, Texas, United States